CLINICAL TRIAL: NCT05228678
Title: Persistent Dyspnea in Post-COVID-19 Patients: Value of Cardiopulmonary Exercise Tests
Brief Title: Persistent Dyspnea in Post COVID_19 and Pulmonary Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Sayed Ali, Assistant lecturer, Assiut University
Other Study IDs: post COVID_19 and dyspnea
Record Dates: First submitted 2022-02-06; First posted 2022-02-08 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: covid_19 Patients
Keywords: post covid_19,dyspnea, cardiopulmonary exercise
MeSH Terms: conditions — Dyspnea | interventions — Exercise Test; Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dyspnea group: Patients with prior diagnosis of COVID-19 and present with persistent dyspnea after 12 weeks of occurrence of symptoms every patient in this group will undergo Cardiopulmonary exercise test (CPET) protocol: -
  1. As regard CPET protocol we prepared incremental treadmill exercise protocol in which the work rate increased at one-minute intervals.
  2. The following parameters observed:
     1. Metabolic response
        * Oxygen consumption VO2 (ml/ min):
        * P ETO2: Is the end-tidal O2 tension as measured from the exhaled air.
        * P ETCO2: Is the end-tidal CO2 tension as measured from the exhaled air. Normally decreased during exercise.
        * Anaerobic Threshold (AT): Is defined as the VO2 (in L/min) at which there is substantial transition to anaerobic metabolism to produce extra energy
     2. Ventilatory response
        * Minute ventilation :
        * Breathing reserve(BR): Breathing reserve = measured/predicted minute ventilation maximum
        * Tidal volume (VT):
        * Respiratory frequency (RF)
  Interventions: Diagnostic Test: cardiopulmonary exercise tests
- Control group: Patients with prior diagnosis of COVID-19, fully recovered, without persistent dyspnea every patient in this group will undergo Cardiopulmonary exercise test (CPET) protocol: -
  1. As regard CPET protocol we prepared incremental treadmill exercise protocol in which the work rate increased at one-minute intervals.
  2. The following parameters observed:
     1. Metabolic response
        * Oxygen consumption VO2 (ml/ min):
        * P ETO2: Is the end-tidal O2 tension as measured from the exhaled air.
        * P ETCO2: Is the end-tidal CO2 tension as measured from the exhaled air. Normally decreased during exercise.
        * Anaerobic Threshold (AT): Is defined as the VO2 (in L/min) at which there is substantial transition to anaerobic metabolism to produce extra energy
     2. Ventilatory response
        * Minute ventilation :
        * Breathing reserve(BR): Breathing reserve = measured/predicted minute ventilation maximum
        * Tidal volume (VT):
        * Respiratory frequency (RF)
  Interventions: Diagnostic Test: cardiopulmonary exercise tests

INTERVENTIONS:
Diagnostic Test: cardiopulmonary exercise tests — Spirometry
  * forced expiratory volume in 1 second (FEV1) % predicted,
  * forced vital capacity (FVC)% predicted,
  * forced expiratory volume in 1 second /forced vital capacity FEV1 /FVC
  Other Names: spirometry

SUMMARY:
COVID-19 has a high spread rate, millions of people have been infected around the world. Patients complained of different symptoms as fever, dry cough and fatigue which is mild in about 80% of cases, but the severity of the case may progress to develop a respiratory distress or respiratory failure, which may require the need for intensive care unit (ICU)

DETAILED DESCRIPTION:
COVID-19 has a high spread rate, millions of people have been infected around the world. Patients complained of different symptoms as fever, dry cough and fatigue which is mild in about 80% of cases, but the severity of the case may progress to develop a respiratory distress or respiratory failure, which may require the need for intensive care unit (ICU) Many patients with mild or severe COVID-19 do not make a full recovery and have a wide range of chronic symptoms for weeks or months after infection.

Post-COVID-19 syndrome is defined by persistent clinical signs and symptoms that appear while or after suffering COVID-19, persist for more than 12 weeks and cannot be explained by an alternative diagnosis.

Dyspnea is one of the most prevalent symptoms in post-covid-19 patients in up to 29% of patients with post COVID-19 syndrome.

Also, persistent dyspnea in post COVID-19 infection is frequent, it is so far, of unknown mechanism. Cardiopulmonary Exercise Test (CPET) is currently the gold standard technique in the differential diagnosis of dyspnea.

Cardiopulmonary exercise testing (CPET) is useful in the assessment of subjects with chronic lung conditions as it may help to: 1) recognize physiological factors limiting exercise (with or without the presence of psychogenic limiting factors); 2) identify these factors as potential therapeutic targets; 3) allow quantification of the level of impairment; 4) assess the effects of an intervention; and 5) provide prognostic information.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or clinically and radiologically highly suspected Covid19-infection
* Symptom duration at least 12 weeks following first occurrence of symptoms
* Patients with dyspnea score 2, 3 and 4 on mMRC
* No other disease that better could explain the symptoms (dyspnea) than Covid-19

Exclusion Criteria:

* Age <18
* pregnant women
* terminally ill patients
* active covid-19 infection
* previous known severe pulmonary or heart disease
* inability to perform pulmonary function or cardiopulmonary exercise tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are diagnosed as post covid_19 who were admittted to isolation unit of Assiut University Hospitals or visit the post covid_19 outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of 1. Aerobic capacity 2. Total Lung Capacity (TLC) | two years
  Aerobic capacity measured as peak oxygen uptake Total lung capacity measured by spirometry

SECONDARY OUTCOMES:
Assessment of Walking capacity | two years
  measured by 6 Minute Walk Test

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Carod-Artal FJ. Post-COVID-19 syndrome: epidemiology, diagnostic criteria and pathogenic mechanisms involved. Rev Neurol. 2021 Jun 1;72(11):384-396. doi: 10.33588/rn.7211.2021230. English, Spanish. PMID 34042167
- [Result] Fernandez-de-Las-Penas C, Palacios-Cena D, Gomez-Mayordomo V, Florencio LL, Cuadrado ML, Plaza-Manzano G, Navarro-Santana M. Prevalence of post-COVID-19 symptoms in hospitalized and non-hospitalized COVID-19 survivors: A systematic review and meta-analysis. Eur J Intern Med. 2021 Oct;92:55-70. doi: 10.1016/j.ejim.2021.06.009. Epub 2021 Jun 16. PMID 34167876
- [Result] Radtke T, Crook S, Kaltsakas G, Louvaris Z, Berton D, Urquhart DS, Kampouras A, Rabinovich RA, Verges S, Kontopidis D, Boyd J, Tonia T, Langer D, De Brandt J, Goertz YMJ, Burtin C, Spruit MA, Braeken DCW, Dacha S, Franssen FME, Laveneziana P, Eber E, Troosters T, Neder JA, Puhan MA, Casaburi R, Vogiatzis I, Hebestreit H. ERS statement on standardisation of cardiopulmonary exercise testing in chronic lung diseases. Eur Respir Rev. 2019 Dec 18;28(154):180101. doi: 10.1183/16000617.0101-2018. Print 2019 Dec 31. PMID 31852745
- [Result] Debeaumont D, Boujibar F, Ferrand-Devouge E, Artaud-Macari E, Tamion F, Gravier FE, Smondack P, Cuvelier A, Muir JF, Alexandre K, Bonnevie T. Cardiopulmonary Exercise Testing to Assess Persistent Symptoms at 6 Months in People With COVID-19 Who Survived Hospitalization: A Pilot Study. Phys Ther. 2021 Jun 1;101(6):pzab099. doi: 10.1093/ptj/pzab099. PMID 33735374